CLINICAL TRIAL: NCT03652350
Title: A Pilot Study to Exam the Flexibility, Safety and Efficacy of Using Microwave Ablation in Patients With Ground Glass Nodules
Brief Title: CT-guided Microwave Ablation in Ground Glass Nodules
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Wuxi People's Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KYLLH2018039
Record Dates: First submitted 2018-08-14; First posted 2018-08-29 (Actual); Last update posted 2018-09-27 (Actual); Status verified 2018-09

CONDITIONS: Ground Glass Nodules Less Than 3cm

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Use CT-guided microwave ablation in Ground Glass Nodules ≤ 3cm (Experimental): Patients with Ground Glass Nodules ≤ 3cm were treated with CT-guided microwave ablation
  Interventions: Procedure: CT-guided microwave ablation

INTERVENTIONS:
Procedure: CT-guided microwave ablation — Using thermal ablation electrode ECO-100AL6 probe target the GGN zone with the guidance performed by CT (Bright Speed Scanner )

SUMMARY:
In order to conduct a multicenter comparative effectiveness clinical research of phase II to investigate safety and efficacy of applying microwave ablation in patients with Great-glass lung nodules ≤ 3cm, a single center, non-randomized, open label pilot study is conducted to examine the flexibility, safety and efficacy of using Microwave Ablation in Patients with Ground Glass Nodules that are poor candidate of surgery.

DETAILED DESCRIPTION:
Lung cancer is the most common cancer worldwide contributing 13% of the total number of new cases diagnosed. The main treatments of lung cancer are based on surgical resection and adjuvant postoperative chemotherapy. However, the patients who are intolerant of surgery wouldn't be benefit from surgical resection. Microwave ablation provide new choice for lung cancer, which can effectively treat early lung cancer. The diagnosis of early lung cancer can be based on the results of biopsy of ground-glass nodules (GGNs), which is one of the diagnostic criteria for preoperative diagnosis of early lung cancer. The microwave ablation is the good choice for patients who cannot tolerate surgical resection. However, the flexibility, safety and efficacy of using Microwave Ablation in Patients with Ground Glass Nodules are still unclear.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent, inclusive of release of medical information.
2. Age ≥ 18 years
3. CT scan indicates presence of Ground Glass Lung Nodules less than 30mm
4. Willing to comply with all protocol required follow-up: 30 days and 90 days post microwave ablation
5. Patients who cannot tolerate surgical resection due to cardiopulmonary dysfunction and advanced age
6. Patients who refuse surgical resection
7. Patients who don't have serious complications

Exclusion Criteria:

1. Unable to give informed consent or potential for noncompliance with the study protocol in the judgement of the investigator
2. Pregnant or breast-feeding at time of screening
3. Active skin infection and ulceration around the percutaneous site
4. Severe pulmonary fibrosis, especially drug-induced pulmonary fibrosis
5. Tendency of severe bleeding, platelets less than 50 × 109 / L and severe blood coagulation disorders. Anticoagulant therapy and/or antiplatelet agents should be discontinued for at least 5d-7d before microwave ablation.
6. Ablation of the ipsilateral malignant pleural effusion is not well controlled
7. Liver, kidney, heart, lung, brain dysfunction, severe anemia, dehydration and serious disorders of nutritional metabolism, cannot be corrected or improved in the short term, severe systemic infection, high fever (> 38.5 oC)
8. Extensive extrapulmonary metastasis, expected to survive < 3 months
9. Eastern Cooperative Oncology Group (ECOG) performance status > 3

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2018-09-13 (Actual); Primary Completion 2019-02 (Estimated); Study Completion 2019-02 (Estimated)

PRIMARY OUTCOMES:
Number of participants recruited; Number of participants complied with protocol; Number of participants finished the study; Number of participants withdrew from the study | 6 months
  Feasibility data that help identify potential population target of CT-guided microwave ablation

SECONDARY OUTCOMES:
Number of participants with treatment-related adverse events assessed by CTCAE v4.0 | 6 months
  Safety data of CT-guided microwave ablation
Number of participants successfully removed ground glass nodules and no relapse in follow-up visit | 6 months
  Efficacy data of CT-guided microwave ablation
Confounding variables identified that interfere with efficacy of microwave ablation | 6 months
  Age, sex, medical history and ground glass nodules size examined by regression analysis

CONTACTS AND LOCATIONS:
Locations (1):
- Wuxi People's Hospital, Wuxi, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Yes